CLINICAL TRIAL: NCT03460782
Title: An Expanded Access Program of Ipilimumab for Patients With Glioblastomas and Gliomas
Status: No longer available | Type: Expanded Access
Sponsor: Center Trials & Treatment (Other)
Collaborators: BioGene Pharmaceutical Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: PST-9-IP
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Glioblastoma; Glioma of Brain
Keywords: Ipilimumab; Glioblastoma; Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Ipilimumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Ipilimumab — Each patient receives Ipilimumab in regimen and dose according to the official manufacturer's instructions (IV 1 mg / kg every 6 weeks for maximum of 4 doses).
  Participation of the patient in the program must necessarily be agreed with the current treatment and contain a written agreement with the attending physician.
  This program is not covered by health insurance. For patients in the postoperative period to provide a mandatory conclusion of histology and molecular-genetic for the identified mutations and the type of tumor.
  Other Names: MDX-010

SUMMARY:
IPILIMUMAB Extended Access Program for patients who received chemotherapy and / or radiation therapy before the protocol, before or after the operation.

DETAILED DESCRIPTION:
It is not yet known which protocols are a better treatment for glioblastoma or glioma.

The ipilimumab extended-access program for patients who received previous chemotherapy and / or radiation therapy by protocol, before ((for non-operable cases) or after the operation.

Monoclonal antibodies of CTLA-4, such as ipilimumab, may block tumor growth in different ways by targeting certain cells and activating the patient's immune system to fight the disease.

ELIGIBILITY:
Inclusion Criteria:

* Glioblastoma.
* Glioma Brain.
* Male or female subjects aged ≥18 years.
* Histopathological evidence of glioblastoma or glioma.
* Patients still alive must provide informed consent if required by local regulations
* Maximal tumor diameter (including residual tumor and resection cavity if subjects had tumor resection rather than only stereotactic biopsy) up to 7cm or less.
* Karnofsky performance status (Appendix 2) of ≥60.
* Availability of a paraffin-embedded or frozen tumor-tissue block with a minimum of 0.5 cm2 and 5 unstained slides from the glioblastoma or glioma tissue specimen.
* Not earlier than 35 days after surgery.
* An interval of at least 2 week for stereotactic biopsy from the start of study treatment.
* A contrast-enhanced MRI must be obtained within 7 days of the first dose of study treatment.
* Adequate hematologic, hepatic, and renal function defined by test
* Women must have a negative serum or urine pregnancy test before 24 hours of initiation of study drug.
* Any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL to be defined as post-menopausal.

Women receiving ipilimumab will be instructed to adhere to contraception for a period of 35 weeks after the last dose of program.

* Men receiving ipilimumab and who are sexually active will be instructed to adhere to contraception for a period of 39 weeks after the last dose of program.
* Contraception is not required for men with documented vasectomy.
* Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.
* Women must not be breastfeeding.
* Willing to and capable of providing written informed consent prior to any program related procedures.
* Ability and willingness to comply scheduled visits, treatment plans, laboratory tests, and other program-related procedures.

Exclusion Criteria:

* Prior systemic treatment anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
* Planned participation in another study intended for therapy of glioma or glioblastoma.
* Primary brainstem or spinal cord tumor.
* Diffuse leptomeningeal gliomatosis.
* Сonfirmed mutation of the IDH1/2 genes.
* Stem or dendritic cell therapy 60 days before the program or 45 days after the last infusion of ipilimumab.
* Systemic treatment with either immunosuppressive doses of corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 21 days of study drug administration.
* Patients on a standard high-dose steroid taper after craniotomy or stereotactic biopsy may have received a higher dose of corticosteroids within 21 days of registration, however must be at a dose < 5 mg daily prednisone or bioequivalent per day within 7 days prior to initiation of study drug.
* Patients requiring adrenal replacement with corticosteroids are eligible if the steroids are at doses ≤ 10 mg prednisone or bioequivalent per day in the absence of active autoimmune disease.
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) are allowed.
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent.
* Prior organ transplantation, including allogeneic stem cell transplantation.
* Known history of, or any evidence of active, non-infectious pneumonitis within the last 5 years.
* Known severe (NCI-CTCAE v4.03 Grade 3 or 4) infusion-related allergy or acute hypersensitivity reaction attributed to any monoclonal antibody, any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
* Unable tolerate an MRI, or have a contraindication to MRI.
* Active infection requiring systemic therapy.
* Positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus (HCV antibody) indicating acute or chronic infection.
* Vaccination within 5 weeks of the first dose of study drug and while on trials is prohibited except for administration of inactivated vaccines.

ATTENTION: Seasonal influenza vaccines for injection are live attenuated vaccines, and are not allowed.

* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ NY Heart Association - CC II), or serious cardiac arrhythmia requiring medication.
* All other unstable, severe, or chronic medical or psychiatric conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis, recent (within the past year) or active suicidal idea in behavior, or laboratory abnormalities that may increase the risk associated with program or judgment of the investigator, would make the patient participation impossible.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- University "Mother Theresa" Hospital Center; Oncology Department, Tirana, Albania
- University Clinical Center of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Complex Oncology Center, Plovdiv, Bulgaria
- Clinical Hospital Osijek; Dept For Oncology & Radiotherapy, Osijek, Croatia
- Institut of Oncology Al. Trestioreanu Bucharest; Oncology, Bucharest, Romania
- Russia (3):
  - Regional Oncology Hospital, Irkutsk
  - Rostov Cancer Research Institute, Rostov-on-Don
  - Primorsky Regional Oncology Center, Vladivostok
- Clinical Hospital Center Bezanijska kosa; Clinic for Oncology, Belgrade, Serbia
- Switzerland (2):
  - Inselspital Bern; Medizinische Onkologie, Bern
  - Stadtspital Triemli; Frauenklinik, Zurich